CLINICAL TRIAL: NCT01735448
Title: Advancing the Understanding of Barriers and Facilitators for Tobacco Prevention, Cessation Treatments, Doctor Visits for Related Illnesses and Health Research for Aboriginal Australians
Brief Title: Improving Health for Aboriginal People Through Tobacco Related Research
Status: Completed | Type: Observational
Sponsor: The Queen Elizabeth Hospital (Other)
Collaborators: University of Adelaide (Other)
Responsible Party: Principal Investigator, Kristin Carson, Senior Scientist, The Queen Elizabeth Hospital
Other Study IDs: 04-12-472; AHREC 04-12-472 (Other: Aboriginal Health Research Ethics Committee)
Record Dates: First submitted 2012-11-23; First posted 2012-11-28 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Tobacco Dependence
Keywords: smoking cessation; tobacco; addiction; Aboriginal; youth; Indigenous; pharmacological; focus group; interview
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Behavior, Addictive | interventions — Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (13):
- Aboriginal smoker, male, Adelaide: Focus group: Aboriginal smoker, male from Adelaide
  Interventions: Other: Focus group; Other: Survey
- Aboriginal smoker, female, Adelaide: Focus group: Aboriginal smoker, female, from Adelaide
  Interventions: Other: Focus group; Other: Survey
- Aboriginal ex/non-smoker, male, Adelaide: Focus group: Aboriginal ex/non-smoker, male, from Adelaide
  Interventions: Other: Focus group; Other: Survey
- Aboriginal ex/non-smoker, female, Adelaide: Focus group: Aboriginal ex/non-smoker, female, from Adelaide
  Interventions: Other: Focus group; Other: Survey
- Healthcare workers, Adelaide: Focus group: Healthcare workers who are based in Adelaide and work with Aboriginal patients
  Interventions: Other: Focus group; Other: Survey
- Healthcare workers, Murray Bridge: Focus group: Healthcare workers who are based in Murray Bridge and work with Aboriginal patients
  Interventions: Other: Focus group; Other: Survey
- Aboriginal smoker, male, Murray Bridge: Focus group: Aboriginal smoker, male, from Murray Bridge
  Interventions: Other: Focus group; Other: Survey
- Aboriginal smoker, female, Murray Bridge: Focus group: Aboriginal smoker, female, from Murray Bridge
  Interventions: Other: Focus group; Other: Survey
- Aboriginal ex/non-smoker, male, Murray Bridge: Focus group: Aboriginal ex/non-smoker, male, from Murray Bridge
  Interventions: Other: Focus group; Other: Survey
- Aboriginal ex/non-smoker, female, Murray Bridge: Focus group: Aboriginal ex/non-smoker, female, from Murray Bridge
  Interventions: Other: Focus group; Other: Survey
- Key community stakeholders: One-on-one interviews with 10 key Aboriginal community stakeholders
  Interventions: Other: One-on-one interviews; Other: Survey
- Respiratory physicians: One-on-one interviews with 10 Respiratory physicians
  Interventions: Other: One-on-one interviews; Other: Survey
- Consultants and General Practitioners: One-on-one interviews with 10 consultants and/or GP's
  Interventions: Other: One-on-one interviews; Other: Survey

INTERVENTIONS:
Other: Focus group — Initially, ten focus groups with an average sample size of 5-7 participants each will be performed in two communities within South Australia, one being Adelaide and the other Murray Bridge, this includes focus groups held with healthcare workers.
  The proposed focus groups will be conducted by experienced mediators who have undertaken Aboriginal cultural awareness training and have experience in qualitative research methods. Both mediators have also been involved in all aspects of project development and consultation with Aboriginal Elders and key stakeholders since its conception.
  We will be using topic guides (reviewed by Aboriginal Elders and researchers) that will be semi-structured with open-ended questions designed to encourage group discussion around smoking cessation and the use of pharmacotherapies in particular, in addition to other objectives identified during the consultation phase of this research.
  Groups: Aboriginal ex/non-smoker, female, Adelaide; Aboriginal ex/non-smoker, female, Murray Bridge; Aboriginal ex/non-smoker, male, Adelaide; Aboriginal ex/non-smoker, male, Murray Bridge; Aboriginal smoker, female, Adelaide; Aboriginal smoker, female, Murray Bridge; Aboriginal smoker, male, Adelaide; Aboriginal smoker, male, Murray Bridge; Healthcare workers, Adelaide; Healthcare workers, Murray Bridge
Other: One-on-one interviews — One-on- one interviews will be held with both medical clinicians and key stakeholders and will be conducted by existing TQEH (The Queen Elizabeth Hospital), Clinical Practice Unit employees, experienced in qualitative research. Informed consent will be required and the interview will be audio taped to allow analysis of the qualitative data. All interviews will remain anonymous, unless the interviewee prefers to be named. In this case, they will be named in the acknowledgement section of all publications and presentations. Moderator guides have been developed and reviewed in the same process undergone by the focus group moderator guides
  Groups: Consultants and General Practitioners; Key community stakeholders; Respiratory physicians
Other: Survey — A four page survey will be administered to all focus group and interview participants in addition to select cohorts including tobacco related special interest groups of the Thoracic Society of Australia and New Zealand (TSANZ). The survey will include demographic data, smoking history and current smoking status (questions related to smoking for current tobacco users include the Fagerstrom test for nicotine dependence, multiple Likert scales for cravings, motivation to quit, confidence etc.) and Likert scales examining perceptions, attitudes and knowledge about tobacco use, cessation, prevention, health and research in the Aboriginal setting.

SUMMARY:
Aim: To identify barriers and facilitators in the uptake of smoking cessation pharmacotherapies, tobacco prevention, doctor visits, smoking amongst youth, community held health priorities and barriers to research in Aboriginal Australians from the perspectives of:

* Aboriginal smokers and ex/non-smokers
* Aboriginal Healthcare workers
* Consultants/general practitioners, and
* Key stakeholders in Aboriginal health

Focus groups, one-on-one interviews and surveys will be conducted to provide information at the 'grass-roots' level including examinations into perceived differences in locally held beliefs, attitudes, knowledge, traditional practices and the cultural and social constructs, to assist implementation of future tobacco cessation/prevention interventions and treatment of smoking related illnesses. This information can be used to improve the health of Aboriginal people by identifying inadequacies in current practices and highlighting what these are through the eyes of community members, healthcare workers, consultants/general practitioners and key stakeholders. We also intend on examining any facilitators that are identified as positive and working aspects of current initiatives e.g. community infrastructure, in an effort to not 'reinvent the wheel' and acknowledge what is working.

DETAILED DESCRIPTION:
We will identify barriers and facilitators for the implementation of smoking cessation pharmacotherapies, tobacco prevention, doctor visits, youth and smoking, community held health priorities and barriers to research through:

1. Multiple focus groups held within 2 communities with Aboriginal smokers and ex/non-smokers, and
2. Focus groups with healthcare workers serving these communities, and
3. Qualitative one-on-one interviews with key stakeholders in Aboriginal communities
4. Qualitative one-on-one interviews with specialists/doctors working with Aboriginal patients
5. Surveys with all participants mentioned above
6. Surveys with specialist groups including members of tobacco related special interest groups of the Thoracic Society of Australia and New Zealand (TSANZ)

Smoking cessation is one of the most important ways to improve the prognosis of patients with respiratory diseases. Despite being over represented in the burden of smoking related morbidity and mortality, very little methodologically rigorous research has been conducted to evaluate and/or enhance the uptake of smoking cessation pharmacotherapies and smoking prevention for Aboriginal Australians, as evident in our two recent (2012) Cochrane meta-analyses and through extensive consultation over the past two years with Aboriginal Elders, key stakeholders, researchers and experts throughout Australia. Moreover, many of the healthcare workers and some doctors on the frontline are reporting that they do not believe they have the skills or ability to offer smoking cessation/prevention initiatives to these patients, and perhaps more importantly, admit to the attitude of 'even if I did, it's not going to work, so why bother'.

In light of this gap in knowledge, our project relates specifically to understanding and improving the lung health of Aboriginal Australians, the cohort with the greatest burden of disease and lowest life expectancy, through qualitative analyses. A total of 10 focus groups, 30 one-on-one interviews and approximately 120 surveys (unless data saturation is reached sooner) will be carried out in collaboration with Aboriginal community involvement. The information obtained from these will provide an overall picture of the barriers and enablers from the perspectives of the various individuals involved, being:

* Aboriginal participants from urban, regional and rural cohorts (8 focus groups plus surveys)
* Aboriginal healthcare workers from urban, regional and rural cohorts (2 focus groups plus surveys)
* Respiratory consultants who see Aboriginal patients (10 one-on-one interviews plus surveys)
* Key stakeholders in Aboriginal health including Aboriginal liaison officers, Aboriginal health councils, Elders & influential figures in communities (10 one-on-one interviews plus surveys)
* Medical Consultants who see Aboriginal patients (2 one-on-one interviews plus surveys from each of the following disciplines: General Practitioners, cardiology, neurology, oncology and vascular; total of 10, or until data saturation)

Triangulation will occur at multiple levels to improve credibility and dependability including: data collection (focus groups, interviews and surveys), investigators (minimum five investigators involved throughout various aspects of the study), data sources (multiple locations, communities and venues), analysis methods (Grounded theory and Triandis model of behavioural change).

In addition a detailed audit trail will be kept and all focus groups and interviews will undergo feedback (confirmation of accuracy and interpretation) by participants. Quasi-statistics will also be employed as part of the analysis methods.

ELIGIBILITY:
Inclusion Criteria:

Male Smokers

* Willing to participate
* Identifies as an Aboriginal person
* Uses more than 10 cigarettes or cigarette equivalent per week
* Has lived in the relevant community for >12 months

Female Smokers

* Willing to participate
* Identifies as an Aboriginal person
* Uses more than 10 cigarettes or cigarette equivalent per week
* Has lived in the relevant community for >12 months

Male Non/Ex Smokers

* Willing to participate
* Identifies as an Aboriginal person
* Has not used tobacco for >3 months
* Has lived in the relevant community for >12 months

Female Non/Ex Smokers

* Willing to participate
* Identifies as an Aboriginal person
* Has not used tobacco for >3 months
* Has lived in the relevant community for >12 months

Healthcare worker

* Willing to participate
* Has provided healthcare to people from Aboriginal people for at least 25% of employment hours over the past 12 months, or
* Has provided healthcare to people from Aboriginal people for at least 5 years of their working career
* Is a qualified healthcare worker

GP's / Specialists

* Willing to participate
* Has provided clinical care to people from Aboriginal people over a 12 month period (at least one consult per week or equivalent)
* Is a qualified General Practitioner or,
* Is a qualified doctor specialising in one of the following disciplines: respiratory, vascular, neurology, oncology, cardiology

Key Stakeholders

* Willing to participate
* Currently working/has worked in Aboriginal health as a primary focus of the position, or
* Is a community Elder, or
* Is influential in Aboriginal health/communities

Exclusion Criteria:

* Cannot speak English
* Cannot sign a consent
* Does not have the intellectual capacity required to respond to questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who agree to be involved in the focus groups will be recruited via existing community contacts (e.g., Aboriginal elders, leaders of community groups and doctors who support the planned research) in urban Adelaide and regional Murray Bridge. We also intend on actively recruiting through clinic visits made by our visiting respiratory clinicians. Copies of the participant information sheet and consent form will be disseminated via local healthcare workers to seek focus group volunteers and via existing contacts in health and by word of mouth for one-on-one interview participants. Survey participants will be recruited as per above methods in addition to use of delegate lists and mail outs.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2013-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Determine the barriers and facilitators to pharmacological initiatives for tobacco cessation in Aboriginal populations | 18 months
  Qualitative analysis (focus groups, one-on-one interviews and surveys). The use of pharmacotherapies for smoking cessation significantly improves the probability of successful abstinence. Identification of the barriers and facilitators for tobacco cessation pharmacotherapies will be determined through these qualitative discussions and mixed method approaches

SECONDARY OUTCOMES:
Determine the barriers and facilitators for tobacco prevention initiatives, particularly related to Aboriginal youth | 18 months
  Qualitative analysis (focus groups, one-on-one interviews and surveys). The use of tobacco prevention initiatives significantly improves the probability of lower tobacco prevalence long-term. Identification of the barriers and facilitators for tobacco prevention initiatives will be determined through these qualitative discussions and mixed method approaches
Identify the barriers and facilitators for doctor visits by Aboriginal people | 18 months
  Qualitative analysis (focus groups, one-on-one interviews and surveys). Regular doctor visits by Aboriginal people can significantly reduce the progression of chronic illnesses, improve quality of life and reduce health care costs. Identification of the barriers and facilitators for these doctor visits, particularly with Respiratory physicians, will be determined through these qualitative discussions and mixed method approaches
Identify barriers and facilitators to research initiatives in Aboriginal people and identify self-reported health priorities | 18 months
  Qualitative analysis (focus groups, one-on-one interviews and surveys). Research in Aboriginal populations are often lengthy and in many cases fail to achieve their objectives, often due to inappropriate methodology or a lack of consultation with Aboriginal Elders or key stakeholders research initiatives particularly related to tobacco and chronic illnesses will be determined through these qualitative discussions and mixed method approaches. In addition, we aim to identify health priorities identified by participants within the focus groups, one-on-one interviews and surveys that can be targeted for future research initiatives.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin V Carson, PhD, Principal Investigator — University of Adelaide; Brian J Smith, MBBS, PhD, Study Director — The Queen Elizabeth Hospital; Adrian J Esterman, PhD,MSc,BSc, Study Director — University of South Australia; Matthew J Peters, MBBS, PhD, Study Director — Concord Hospital
Locations (3):
- Australia (3):
  - The Basil Hetzel Institute for Translational Health Research, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - Murray Mallee Community Health Service; Aboriginal Primary Health Care Unit, Murray Bridge, South Australia

IPD SHARING:
Plan to Share IPD: Yes
Available on request

REFERENCES:
- [Background] Carson KV, Brinn MP, Labiszewski NA, Peters M, Chang AB, Veale A, Esterman AJ, Smith BJ. Interventions for tobacco use prevention in Indigenous youth. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD009325. doi: 10.1002/14651858.CD009325.pub2. PMID 22895988 (Retraction: PMID 34847239 Cochrane Database Syst Rev. 2021 Nov 30;11:CD009325)
- [Background] Carson KV, Brinn MP, Peters M, Veale A, Esterman AJ, Smith BJ. Interventions for smoking cessation in Indigenous populations. Cochrane Database Syst Rev. 2012 Jan 18;1:CD009046. doi: 10.1002/14651858.CD009046.pub2. PMID 22258998